CLINICAL TRIAL: NCT01231555
Title: Phase 2b Study to Select a Once Daily Oral Dose of GSK2248761 Administered With Tenofovir/Emtricitabine or Abacavir/Lamivudine in HIV-1 Infected Antiretroviral Therapy Naive Adult Subjects
Brief Title: Dose-finding Study of GSK2248761 in Antiretroviral Therapy-Naive Subjects (SIGNET)
Acronym: SIGNET
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113404
Record Dates: First submitted 2010-10-14; First posted 2010-11-01 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-08

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: antiretroviral; HAART; NNRTI; emtricitabine; Sexually Transmitted Disease; antiretroviral therapy (ART)-naive adults; Immunologic Deficiency Syndrome; tenofovir; abacavir; Retroviridae Infections; GSK2248761; lamivudine; Acquired ImmunoDeficiency Syndrome (AIDS); HIV infection; efavirenz
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; Immunologic Deficiency Syndromes; Retroviridae Infections; HIV Infections | interventions — IDX 899; efavirenz

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GSK2248761 100 mg once daily (Experimental): In combination with either abacavir/lamivudine FDC qd or tenofovir/emtricitabine FDC qd
  Interventions: Drug: GSK2248761 100 mg once daily
- GSK2248761 200 mg once daily (Experimental): In combination with either abacavir/lamivudine FDC qd or tenofovir/emtricitabine FDC qd
  Interventions: Drug: GSK2248761 200 mg once daily
- Efavirenz 600 mg once daily (Active Comparator): In combination with either abacavir/lamivudine FDC qd or tenofovir/emtricitabine FDC qd
  Interventions: Drug: Efavirenz 600 mg once daily

INTERVENTIONS:
Drug: GSK2248761 100 mg once daily — 1x100 mg capsule plus matching placebo
  Arms: GSK2248761 100 mg once daily
Drug: GSK2248761 200 mg once daily — 2x100 mg capsules
  Arms: GSK2248761 200 mg once daily
Drug: Efavirenz 600 mg once daily — 1x600mg tablet
  Arms: Efavirenz 600 mg once daily

SUMMARY:
This 96 week, Phase 2b study in 150 HIV-1 infected antiretroviral (ART) naive adult subjects consists of a dose-ranging evaluation of GSK2248761 at blinded doses of 100 mg and 200 mg once daily with a control arm of open-label efavirenz (EFV) 600 mg once daily. The background ART for all 3 arms will be chosen by the Investigators and will be either abacavir/lamivudine [ABC/3TC] or tenofovir/emtricitabine [TDF/FTC] fixed dose combination (FDC) tablets. Antiviral activity, safety, PK, and development of viral resistance will be evaluated.

DETAILED DESCRIPTION:
Study SGN113404 is a phase 2b randomized, partially blinded, multicenter, parallel group, dose-ranging study. The study will be conducted in approximately 150 HIV-1 infected ART naïve subjects. The background NRTIs to be co-administered with GSK2248761 or EFV will be selected by Investigators prior to randomization and will be either abacavir/lamivudine (ABC/3TC) or tenofovir/emtricitabine (TDF/FTC) fixed dose combination (FDC) tablets.

Subjects will participate in a Screening period (Day -28 to Day -1). Subjects may be re-screened once. Subjects will be randomized 1:1:1 to receive 100 mg of GSK2248761 once daily (50 subjects), 200 mg of GSK2248761 once daily (50 subjects) or 600 mg of EFV once daily (50 subjects). All three arms will be combined with either 300 mg/200 mg TDF/FTC or 600 mg/300 mg ABC/3TC, as chosen by the Investigator. The Investigators and subjects will be blinded to the dose of GSK2248761 being administered but will know whether they receive EFV or GSK2248761. The randomization will be stratified by HIV-1 viral load (VL) at screening, < 100,000 copies/mL or >/ 100,000 copies/mL as well as the choice of backbone NRTI, TDF/FTC or ABC/3TC.

This study will be enrolled in two stages. The first stage of the study will enroll approximately 30 subjects, at which time enrollment will be paused. An analysis of safety and tolerability will be reviewed by a safety review committee (SRC) once all subjects enrolled in Stage 1 reach Week 4. The SRC review will determine if the safety and tolerability profile of GSK2248761 supports the continuation of the trial and enrollment of an additional 120 subjects. All subjects will continue on study medications during this Week 4 analysis.

Additional analyses will be conducted once all subjects complete Week 4, Week 16, Week 24 and Week 48. A second review of the safety and tolerability of GSK2248761 will be performed by the SRC once all subjects reach Week 4. There will not be a pause in the study during the Week 4 analysis of all subjects.

The Week 16 and Week 24 analyses will be used respectively to select and confirm the optimal dose of GSK2248761 for continuation. This dose will be selected based on a statistical analysis of antiviral activity, safety and tolerability criteria. If, after confirmation of the optimal dose of GSK2248761 by the Week 24 analysis, both doses are considered acceptable based on efficacy, safety and PK data, then both arms will be continued through Week 48.

Beyond Week 48, those subjects who were randomized to the non-selected dose of GSK2248761 and have not met any criteria for discontinuation will be given the option to switch to the selected dose of GSK2248761 or to discontinue permanently from the study. Once they have switched to the selected dose they will be in the Open-Label phase of the study through Week 96. After Week 96, subjects receiving GSK2248761 will be given the option to continue to receive GSK2248761 until it is locally approved and commercially available, as long as they continue to derive clinical benefit without a protocol-defined reason for discontinuation.

Subjects randomized to EFV will have the option to continue to receive EFV through Week 96 unless they meet a protocol-defined reason for discontinuation. All subjects will have the option to continue TDF/FTC or ABC/3TC through Week 96. After Week 96, subjects will be expected to obtain local access to all commercially available ART.

Randomization will be stratified by:

* HIV-1 RNA < or >/ 100,000 copies/mL at screening
* Use of ABC/3TC or TDF/FTC FDC tablets as initial background ART

Switch of a background NRTI for toxicity management to an alternative marketed NRTI is allowed once. Switches of a background NRTI for any other reason are not permitted in the study. A switch of GSK2248761 or EFV is not allowed.

Study Endpoints /Assessments: Subjects will have assessments performed which will include baseline demographics, disease characteristics, and safety (laboratory and clinical evaluations). On study safety, efficacy, virologic, immunologic, and PK evaluations will be conducted.

Primary Endpoint: The proportion of subjects with HIV-1 RNA <50copies/mL at Week 16. Dose selection will be based primarily on antiviral activity and tolerability in conjunction with immunologic, safety, virologic resistance and PK measures. Data from the Week 24 analysis will be used to confirm dose selection.

ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected adults greater than or equal to 18 years of age. A female is eligible to enter and participate in the study if she is (1) Non-childbearing potential, (2) Child-bearing potential, with a negative pregnancy test at screen and Day 1 and agrees to use protocol-specified methods of birth control while on study
* HIV-1 infection with a screening plasma HIV-1 RNA greater than or equal to 1000 copies/mL
* CD4+ cell count greater than or equal to 200 cells/mm3
* Antiretroviral-naive

Exclusion Criteria:

* Any pre-existing physical or mental condition (including substance abuse disorder) which, in the opinion of the Investigator, may interfere with the subject's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the subject
* Any condition which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the drug or render the subject unable to take oral medication
* Women who are currently breastfeeding
* Any evidence of an active Centers for Disease and Prevention Control (CDC) Category C disease [CDC,1993], except cutaneous Kaposi's sarcoma not requiring systemic therapy
* History of ongoing or clinically relevant hepatitis within the previous 6 months, including chronic hepatitis B virus (HBV) infection (HBsAg positive). Asymptomatic individuals with chronic hepatitis C virus (HCV) infection will not be excluded, however Investigators must carefully assess if therapy specific for HCV infection is required; subjects who are anticipated to require such therapy during the randomized portion of the study must be excluded
* History of liver cirrhosis with or without hepatitis viral co-infection
* Ongoing or clinically relevant pancreatitis
* History of the following cardiac diseases: myocardial infarction, congestive heart failure, documented hypertrophic cardiomyopathy, sustained ventricular tachycardia
* Personal or known family history of prolonged QT syndrome
* History or presence of allergy or intolerance to the study drugs or their components, or a history of drug or other allergy that, in the opinion of the Principal Investigator, contraindicates their participation. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled
* Evidence of viral resistance to any antiviral drug indicative of primary transmitted resistance in a screening or historical resistance test result
* Any acute laboratory abnormality at screening, which, in the opinion of the Investigator, would preclude the subject's participation in the study of an investigational compound. Any verified Grade 4 laboratory abnormality at screening would exclude a subject from study participation unless the Investigator can provide a compelling explanation for the laboratory result(s) and has the assent of the Medical Monitor
* Any of the following laboratory values at screening: (1) Creatinine clearance <50 mL/min via Cockroft-Gault method, (2) Alanine aminotransferase (ALT) greater than or equal to 5 times upper limits of normal (ULN). Subjects with ALT > 2x ULN but <5xULN may participate in the study, if in the opinion of the Investigator and GSK Medical Monitor the lab abnormality will not interfere with the study procedures or compromise subject safety, (3) Alanine aminotransferase (ALT) greater than or equal to 3xULN and bilirubin greater than or equal to 1.5xULN (with >35% direct bilirubin)
* Any clinically significant finding on screening ECG, specifically (a single repeat is allowed to determine eligibility): (1) Heart rate <45 and >100 beats per minute (bpm) (males); <50 and >100 bpm (females). Note: A heart rate from 100 to 110 bpm can be rechecked within 30 minutes to verify eligibility, (2) QRS duration > 120 msec, (3) QTc interval > 450 msec (4) Non-sustained (greater than or equal to 3 consecutive beats) or sustained ventricular tachycardia, (5) Sinus pauses > 2.5 seconds, (6) 2nd degree (Type II) or higher AV (Atrioventricular) block, (7) Evidence of WPW (Wolff- Parkinson-White) syndrome (ventricular preexcitation), (8) Pathologic Q waves (defined as Q wave > 40 msec OR depth >0.4 mV (9) Any other abnormality which in the opinion of the Investigator would interfere with the safety of the subject
* Treatment with any of the following agents within 28 days prior to screening, or has an anticipated need for these agents during the study (1) Radiation therapy or cytotoxic chemotherapeutic agents, (2) Immunomodulators (such as systemic corticosteroids, interleukins, or interferons) Note: Subjects using short-term (<7 day) steroid tapers and inhaled corticosteroids are eligible for enrollment (3) Any non-protocol-specified agent with documented activity against HIV 1 in vitro
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days prior to screening
* Receipt of an experimental drug and/or vaccine within 28 days or 5 half-lives, or twice the duration of the biological effect of the experimental drug or vaccine, whichever is longer, prior to screening
* Immunization within 28 days prior to first dose of IP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-11-18 (Actual); Primary Completion 2011-07-04 (Actual); Study Completion 2011-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (11):
- France (4):
  - GSK Investigational Site, Levallois-Perret
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
- Germany (4):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Spain (3):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Marid

REFERENCES:
- [Background] 1993 revised classification system for HIV infection and expanded surveillance case definition for AIDS among adolescents and adults. MMWR Recomm Rep. 1992 Dec 18;41(RR-17):1-19. PMID 1361652

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 18 November 2010 to 04 July 2011. A total of 150 human immunodeficiency virus (HIV)-1 infected adult participants naïve to antiretroviral therapy (ART) were planned to be enrolled.
Pre-assignment Details: Enrollment was terminated prematurely due to safety findings. At the time of enrollment termination, 23 participants were enrolled who continued into this study. At least 5 interim analyses were planned up to Week 48, however, the study was terminated prior to any of these analyses being conducted.
Groups:
- GSK2248761 100 mg Once Daily: Eligible participants were planned to receive oral GSK2248761 100 milligrams (mg) capsule once daily and matching GSK2248761 Placebo capsule once daily up to 48 weeks, however, participants received GSK2248761 100 mg once daily and matching GSK2248761 Placebo capsule once daily up to 8 weeks due to early termination. All participants received antiretroviral therapy (ART) of Tenofovir disoproxil fumarate/ Emtricitabine (TDF/FTC) 300 mg/200 mg or Abacavir/ Lamivudine (ABC/3TC) 600 mg/300 mg along with the study drug.
- GSK2248761 200 mg Once Daily: Eligible participants were planned to receive oral GSK2248761 200 mg (2x100 mg) capsule once daily up to 48 weeks, however, participants received GSK2248761 200 mg oral capsule once daily up to 8 weeks due early termination. All participants received ART of TDF/FTC 300 mg/200 mg or ABC/3TC 600 mg/300 mg along with the study drug.
- EFV 600 mg Once Daily: Eligible participants were planned to receive oral Efavirenz (EFV) 600 mg tablet once daily up to 48 weeks, however participants received EFV 600 mg tablet once daily up to 16 weeks due to early termination. All participants received ART of TDF/FTC 300 mg/200 mg or ABC/3TC 600 mg/300 mg along with the study drug.
Period: Overall Study
Arm/Group | GSK2248761 100 mg Once Daily | GSK2248761 200 mg Once Daily | EFV 600 mg Once Daily
Started | 8 | 7 | 8
Completed | 0 | 0 | 0
Not Completed | 8 | 7 | 8
Not completed — Study terminated | 8 | 5 | 8
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- GSK2248761 100 mg Once Daily: Eligible participants were planned to receive oral GSK2248761 100 mg capsule once daily and matching GSK2248761 Placebo capsule once daily up to 48 weeks, however, participants received GSK2248761 100 once daily and matching GSK2248761 Placebo capsule once daily up to 8 weeks due to early termination. All participants received ART of TDF/FTC 300 mg/200 mg or ABC/3TC 600 mg/300 mg along with the study drug.
- EFV 600 mg Once Daily: Eligible participants were planned to receive oral EFV 600 mg tablet once daily up to 48 weeks, however participants received EFV 600 mg tablet once daily up to 16 weeks due to early termination. All participants received ART of TDF/FTC 300 mg/200 mg or ABC/3TC 600 mg/300 mg along with the study drug.
- Total: Total of all reporting groups
Arm/Group | GSK2248761 100 mg Once Daily | GSK2248761 200 mg Once Daily | EFV 600 mg Once Daily | Total
Number analyzed (Participants) | 8 | 7 | 8 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.8 (8.01) | 35.9 (6.47) | 35.9 (7.97) | 36.9 (7.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1
  Male | 8 | 6 | 8 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 7 | 7 | 8 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Plasma HIV-1 RNA Below 50 Copies/mL as a Function of Viral Load
Description: This analysis was based on the Missing, Switch or Discontinuation equals Failure (MSDF) algorithm (as codified by the FDA's "snapshot" algorithm) and was adjusted for stratification factors and stage of recruitment. Dose selection was based primarily on antiviral activity and tolerability in conjunction with immunologic, safety, virologic resistance and pharmacokinetic (PK) measures. The efficacy decision criteria was based on an observed difference of >=8% between the two GSK2248761 dosage arms.
Time Frame: Up to Week 16
Population: Intent to treat exposed (ITT-E) population included all randomized participants who received at least one dose of study drug. Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm due to early termination. Only those participants available at indicated timepoints were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2248761 100 mg Once Daily | GSK2248761 200 mg Once Daily | EFV 600 mg Once Daily
Number analyzed (Participants) | 8 | 7 | 8
Participants
  Before switch, Week 4: number analyzed (Participants) | 5 | 4 | 8
  Before switch, Week 4 | 1 | 0 | 3
  Before switch, Week 8: number analyzed (Participants) | 0 | 1 | 8
  Before switch, Week 8 |  | 1 | 3
  Before switch, Week 12: number analyzed (Participants) | 0 | 0 | 4
  Before switch, Week 12 |  |  | 2
  After switch, Baseline switch: number analyzed (Participants) | 6 | 3 | 0
  After switch, Baseline switch | 1 | 1 |
  After switch, Week 1: number analyzed (Participants) | 6 | 5 | 0
  After switch, Week 1 | 3 | 1 |
  After switch, Week 2: number analyzed (Participants) | 8 | 5 | 0
  After switch, Week 2 | 3 | 1 |
  After switch, Week 4: number analyzed (Participants) | 6 | 5 | 0
  After switch, Week 4 | 2 | 1 |

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Adverse Events (AEs)
Description: Adverse event (AE) is an unfavorable change in the health of a participant, including abnormal laboratory findings, that happens during a clinical study or within a certain time period after the study has ended. This change may or may not be caused by the intervention being studied. Serious adverse event (SAE) is an adverse event that results in death, is life-threatening, requires inpatient hospitalization or extends a current hospital stay, results in an ongoing or significant incapacity or interferes substantially with normal life functions, or causes a congenital anomaly or birth defect. Medical events that do not result in death, are not life-threatening, or do not require hospitalization may be considered serious adverse events if they put the participant in danger or require medical or surgical intervention to prevent one of the results listed above.
Time Frame: Up to 20 Weeks
Population: Safety population included all randomized participants who were exposed to the study drug(s) with the exception of any participant with documented evidence of not having consumed any amount of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2248761 100 mg Once Daily | GSK2248761 200 mg Once Daily | EFV 600 mg Once Daily
Number analyzed (Participants) | 8 | 7 | 8
Participants
  Any SAE | 1 | 0 | 1
  Any AE | 8 | 5 | 8

3. Secondary Outcome: Change From Baseline (Day 1) in Plasma HIV-1 RNA Over Period
Description: For summaries and analyses which use HIV-1 RNA level as a continuous measure, the logarithm to base 10 of the value was used. In cases where a sample was retested, the retest value was used. Baseline was defined as the value recorded on Day 1. Change from Baseline is the value at indicated time point minus the Baseline value. Data for participants prior to switch and after the switch has been presented.
Time Frame: Baseline (Day 1) up to Week 16
Population: ITT-E population. Data for only those participants available at the indicated time points were collected and analyzed. Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm due to early termination.
Measure: Mean (Standard Deviation); unit: log10 copies per milliliter
Arm/Group | GSK2248761 100 mg Once Daily | GSK2248761 200 mg Once Daily | EFV 600 mg Once Daily
Number analyzed (Participants) | 8 | 7 | 8
log10 copies per milliliter
  Before switch, Week 2: number analyzed (Participants) | 8 | 5 | 8
  Before switch, Week 2 | -1.863 (0.3496) | -2.018 (0.3427) | -2.131 (0.2818)
  Before switch, Week 4: number analyzed (Participants) | 5 | 4 | 8
  Before switch, Week 4 | -2.140 (0.4528) | -2.134 (0.3055) | -2.334 (0.3384)
  Before switch, Week 8: number analyzed (Participants) | 0 | 1 | 8
  Before switch, Week 8 |  | -2.712 (NA) — Only one participant was analyzed. | -2.723 (0.2411)
  Before switch, Week 12: number analyzed (Participants) | 0 | 0 | 4
  Before switch, Week 12 |  |  | -2.866 (0.2909)
  Baseline switch: number analyzed (Participants) | 6 | 3 | 0
  Baseline switch | -2.046 (0.4943) | -2.170 (0.4990) |
  After switch, Week 1: number analyzed (Participants) | 6 | 5 | 0
  After switch, Week 1 | -2.218 (0.5211) | -2.287 (0.4812) |
  After switch, Week 2: number analyzed (Participants) | 8 | 5 | 0
  After switch, Week 2 | -2.307 (0.4219) | -2.235 (0.3383) |
  After switch, Week 4: number analyzed (Participants) | 6 | 5 | 0
  After switch, Week 4 | -2.380 (0.2749) | -2.482 (0.2567) |

4. Secondary Outcome: Number of Participants With HIV Associated Conditions
Description: HIV associated condition included recurrence of previous conditions. Centre for disease control (CDC) associated conditions and non-CDC associated conditions were planned to be monitored.
Time Frame: Up to 20 Weeks
Population: ITT-E population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2248761 100 mg Once Daily | GSK2248761 200 mg Once Daily | EFV 600 mg Once Daily
Number analyzed (Participants) | 8 | 7 | 8
Participants | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With HIV Disease Progression
Description: Number of participants acquiring clinical disease progression or death during the treatment period were presented. Clinical disease progression was defined as the progression from Baseline (Day 1) HIV disease status in either of these categories; CDC Category A at baseline to CDC Category B event, CDC Category A at baseline to CDC Category C event, CDC Category B at baseline to CDC Category C event, CDC Category C at baseline to new CDC Category C event, CDC Category A, B or C at baseline to death. If no change occurs, it was termed as no disease progression.
Time Frame: Up to 20 Weeks
Population: ITT-E population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2248761 100 mg Once Daily | GSK2248761 200 mg Once Daily | EFV 600 mg Once Daily
Number analyzed (Participants) | 8 | 7 | 8
Participants | 0 | 0 | 0

6. Secondary Outcome: Number of Participants Discontinuing the Study Drugs Due to AEs
Description: Adverse event (AE) is an unfavorable change in the health of a participant, including abnormal laboratory findings, that happens during a clinical study or within a certain time period after the study has ended. This change may or may not be caused by the intervention being studied. Number of participants quitting/ prematurely discontinuing the use of study drug(s) were recorded.
Time Frame: Up to 20 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2248761 100 mg Once Daily | GSK2248761 200 mg Once Daily | EFV 600 mg Once Daily
Number analyzed (Participants) | 8 | 7 | 8
Participants | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Changes in Electrocardiogram (ECG) From Baseline (Day 1) Over 16 Weeks
Description: The QTc interval was assessed by two methods Bazzette's method (QTc[b]) and Federica's method (QTc[f]). Baseline value was recorded at Day 1. Change from Baseline is the value at indicated time point minus the Baseline value. Change from Baseline values were categorized into <30 milliseconds (msec), >=30 but <60 msec, and >=60 msec. The data has been presented for QTcB and QTcF for participants prior to switching the therapy.
Time Frame: Baseline (Day 1) to 16 weeks
Population: Safety population. Data for only those participants available at the indicated time points were collected and analyzed. Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm due to early termination.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2248761 100 mg Once Daily | GSK2248761 200 mg Once Daily | EFV 600 mg Once Daily
Number analyzed (Participants) | 8 | 7 | 8
Participants
  QTcB, Week 2, <30 msec: number analyzed (Participants) | 6 | 5 | 8
  QTcB, Week 2, <30 msec | 6 | 5 | 7
  QTcB, Week 2, >=30 to <60 msec: number analyzed (Participants) | 6 | 5 | 8
  QTcB, Week 2, >=30 to <60 msec | 0 | 0 | 1
  QTcB, Week 4, <30 msec: number analyzed (Participants) | 4 | 4 | 6
  QTcB, Week 4, <30 msec | 4 | 4 | 6
  QTcB, Week 12, <30 msec: number analyzed (Participants) | 0 | 0 | 3
  QTcB, Week 12, <30 msec |  |  | 3
  QTcF, Week 2, <30 msec: number analyzed (Participants) | 6 | 5 | 8
  QTcF, Week 2, <30 msec | 6 | 5 | 8
  QTcF, Week 4, <30 msec: number analyzed (Participants) | 4 | 4 | 6
  QTcF, Week 4, <30 msec | 4 | 4 | 6
  QTcF, Week 12, <30 msec: number analyzed (Participants) | 0 | 0 | 3
  QTcF, Week 12, <30 msec |  |  | 2
  QTcF, Week 12, >=30 to <60: number analyzed (Participants) | 0 | 0 | 3
  QTcF, Week 12, >=30 to <60 |  |  | 1

8. Secondary Outcome: Minimum and Maximum Plasma GSK2248761 Concentration at Week 2
Description: Maximum observed plasma concentration and minimum observed plasma concentration of GSK2248761 was recorded on Week 2. The PK parameters were calculated by standard non-compartmental analysis according to current working practices and using WinNonlin Pro 4.1 or higher. Log transformed values have been presented.
  All calculations of non-compartmental parameters were based on actual sampling times.
Time Frame: At Week 2
Population: The PK Concentration Population included all participants who received GSK2248761, underwent intensive and/or limited PK sampling during the study, and provided evaluable GSK2248761 plasma concentration data. Only the participants available at the time of assessment were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter
Arm/Group | GSK2248761 100 mg Once Daily | GSK2248761 200 mg Once Daily | EFV 600 mg Once Daily
Number analyzed (Participants) | 8 | 7 | 0
micrograms per milliliter
  Cmin: number analyzed (Participants) | 7 | 5 | 0
  Cmin | 0.15 (149) | 0.49 (164) |
  Cmax: number analyzed (Participants) | 4 | 4 | 0
  Cmax | 1.78 (39) | 3.70 (40) |

ADVERSE EVENTS:
Time Frame: Up to 20 weeks
Description: AE (SAE and nSAE) were collected and have been reported for safety population
Arm/Group | GSK2248761 100 mg Once Daily | GSK2248761 200 mg Once Daily | EFV 600 mg Once Daily
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/7 | 1/8
Other Adverse Events (participants affected / at risk) | 8/8 | 5/7 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2248761 100 mg Once Daily (N=8) | GSK2248761 200 mg Once Daily (N=7) | EFV 600 mg Once Daily (N=8)
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2248761 100 mg Once Daily (N=8) | GSK2248761 200 mg Once Daily (N=7) | EFV 600 mg Once Daily (N=8)
Dizziness (Nervous system disorders) | 1 | 0 | 6
Somnolence (Nervous system disorders) | 2 | 2 | 0
Headache (Nervous system disorders) | 0 | 2 | 0
Circadian rhythm sleep disorder (Nervous system disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 3
Bronchitis (Infections and infestations) | 0 | 2 | 1
Anogenital warts (Infections and infestations) | 0 | 0 | 2
Rhinitis (Infections and infestations) | 1 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1
Anal chlamydia infection (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Syphilis (Infections and infestations) | 1 | 0 | 0
Nightmare (Psychiatric disorders) | 2 | 3 | 3
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 0 | 2
Fatigue (General disorders) | 1 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0
Feeling abnormal (General disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Blindness (Eye disorders) | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Palpitations (Cardiac disorders) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.